CLINICAL TRIAL: NCT02945215
Title: A Multicenter, Randomized, Double-blinded, Parallel Controlled Study to Assess the Pharmacokinetics and Safety of Recombinant Human Murine Chimeric Anti CD20 Monoclonal Antibody Injection (IBI301) Compared to Rituximab Injection in CD20 Positive B Cell Lymphoma Patients
Brief Title: A Study to Assess the Pharmacokinetics and Safety of Recombinant Human Murine Chimeric Anti CD20 Monoclonal Antibody Injection (IBI301) Compared to Rituximab Injection in CD20 Positive B Cell Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI301A201
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-06

CONDITIONS: B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBI301 (Experimental)
  Interventions: Drug: IBI301
- Rituximab (Active Comparator)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: IBI301 — IBI301 375mg/㎡
  Arms: IBI301
Drug: Rituximab — Rituximab 375mg/㎡
  Arms: Rituximab

SUMMARY:
Randomised, double-blind, parallel group study to compare PK and PD profiles between IBI301 and rituximab in patients with CD20+ B-cell Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. CD20-positive B-cell lymphoma.
2. 18 years to 65 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Signed an informed consent.
5. Obtained CR (complete remission) or CRu (uncertain complete remission) after the prior therapy.

Exclusion Criteria:

1. Participation in another interventional clinical trial in the past 28 days.
2. Known allergic reactions against monoclonal antibody or rituximab.
3. Rituximab and other anti-CD20 monoclonal antibody used in the past 4 months.
4. Blood concentration of Rituximab>24ug/ml.
5. HIV positive patients.
6. HCV antigen and antibody positive.
7. Acute and chronic hepatitis B virus infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
AUC0-inf of IBI301 and rituximab | 91 days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 91 days
Percentage and absolute value of CD19+ | 91 days
Percentage and absolute value of CD20+ B-cell | 91 days
Positive rate of ADA | 91 days
Positive rate of NAb | 91 days
Safety profiles | up to 1 year
  Including AE type、incidence rate、severity and drug- related
Area under the plasma concentration versus time curve (AUC) | 91days
AUC（0-t） of IBI301 and rituximab | 91 days

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Chinese Academy of Medical Sciences
Locations (12):
- China (12):
  - Beijing cancer hospital, Beijing, Beijing Municipality
  - Peking University third hospital, Beijing, Beijing Municipality
  - The 307th Hospital of Military Medical Sciences, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu province people's hospital, Nanjing, Jiangsu
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No